CLINICAL TRIAL: NCT01162148
Title: Pulmonary Rehabilitation and Inspiratory Muscle Training (IMT) for Patients Following Lung Transplantation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Rabin Medical Center (Other)
Responsible Party: Prof Mordechai R. Kramer M.D, Rabin Medical center, Beilinson Hospital Petach Tikva, 49100 Israel
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: rab581710ctil
Record Dates: First submitted 2010-06-21; First posted 2010-07-14 (Estimated); Last update posted 2010-07-14 (Estimated); Status verified 2010-06

CONDITIONS: Lung Transplantation
Keywords: inspiratory muscle training; pulmonary rehabilitation
MeSH Terms: interventions — Congresses as Topic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1 (Experimental): conventional
  Interventions: Behavioral: Conventional or regular pulmonary rehabilitation program alone
- 2 (Experimental): sham IMT
  Interventions: Device: very low load IMT (sham IMT) alone
- 3 (Experimental): Conventional plus threshold IMT
  Interventions: Device: Conventional or regular pulmonary rehabilitation program + targeted inspiratory resistive or threshold IMT
- 4 (Experimental): threshold IMT alone
  Interventions: Device: Targeted inspiratory resistive or threshold IMT alone

INTERVENTIONS:
Behavioral: Conventional or regular pulmonary rehabilitation program alone — Conventional or regular pulmonary rehabilitation program alone
  Arms: 1
Device: very low load IMT (sham IMT) alone — very low load IMT (sham IMT) alone
  Arms: 2
Device: Conventional or regular pulmonary rehabilitation program + targeted inspiratory resistive or threshold IMT — Conventional or regular pulmonary rehabilitation program + targeted inspiratory resistive or threshold IMT
  Arms: 3
Device: Targeted inspiratory resistive or threshold IMT alone — Targeted inspiratory resistive or threshold IMT alone
  Arms: 4

SUMMARY:
Lung transplantation (LT) is now an established treatment option for patients with a wide variety of end-stage lung diseases- aims to improve quality of life and survival. Pulmonary rehabilitation (PR) is widely recognized as an important component of care of patients with chronic obstructive pulmonary disease (COPD), it improves dyspnea, exercise tolerance, quality of life, and reduces healthcare resource utilization.

The goal of pulmonary rehabilitation following lung transplantation is to enhance the physiological and functional benefits resulting from surgery. Inspiratory muscle Training (IMT) is defined as any intervention with the goal of training the inspiratory muscles. IMT can improve inspiratory muscles strength, endurance and exercise capacity in adults with COPD. IMT provides additional benefits to patients undergoing PR program and is worthwhile even in patients who have already undergone a general exercise reconditioning (GER) program. IMT will provide additional benefits (together or without) PR to patients following lung transplantation. No formal guidelines exist regarding the optimal methods of exercise training component of pulmonary rehabilitation for patients recovering from lung transplantation. This study will evaluate the unique influence of IMT in Patients Following Lung Transplantation.

DETAILED DESCRIPTION:
The post lung transplant patients will participate in a rehabilitation program for 6 months. Participants in the proposed study will belong to one of four intervention groups:

1. Conventional or regular pulmonary rehabilitation program alone(an exercise program that consist 3 main components: aerobic conditioning, resistance training, and flexibility exercises).
2. Very low load IMT(sham IMT) alone.
3. Conventional or regular pulmonary rehabilitation program + Targeted inspiratory resistive or threshold IMT.
4. Targeted inspiratory resistive or threshold IMT alone.

ELIGIBILITY:
Inclusion Criteria:

* Post lung transplant patients attending the pulmonary Institute , will be invited to participate,They will be co-operative and able to perform spirometry; and other lung tests.
* Patients will be stable clinically,for at least one month,the patients will be all new to an IMT program.

Exclusion Criteria:

* Patients with cardiac disease,poor compliance,or requirement of supplemental oxygen.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2010-09; Primary Completion 2010-12 (Estimated); Study Completion 2011-09 (Estimated)

PRIMARY OUTCOMES:
maximal exercise capacity | 9 months after starting interventions
  at 9 months after starting interventions

SECONDARY OUTCOMES:
Lung function (FEV1, FVC) | 9 months after starting interventions
  9 months after starting interventions

CONTACTS AND LOCATIONS:
Overall Officials: Mordechai R Kramer, MD, Principal Investigator — Rabin Medical center, Beilinson Hospital Petach Tikva, 49100 Israel
Locations (1):
- Pulmonary Institute Rabin Medical center, Beilinson Hospital, Petah Tikva, Israel

REFERENCES:
- [Derived] Gutierrez-Arias R, Martinez-Zapata MJ, Gaete-Mahn MC, Osorio D, Bustos L, Melo Tanner J, Hidalgo R, Seron P. Exercise training for adult lung transplant recipients. Cochrane Database Syst Rev. 2021 Jul 20;7(7):CD012307. doi: 10.1002/14651858.CD012307.pub2. PMID 34282853